CLINICAL TRIAL: NCT06803979
Title: The Impact of Delivery Method on the Performance of Elite Athletes.
Brief Title: Impact of Delivery Method Elite Athletes.
Acronym: IDEA
Status: Recruiting | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jan Zapletal, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Other Study IDs: EK-VP/53/2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Delivery; Performance; Caesarean Section; Pregnancy; Athletes
Keywords: delivery; performance; caesarean section; pregnancy; athletes; women health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retires elite athletes: Elite athletes with finished sport career
- Elite athletes currently performing sport: Current elite athletes who are still doing sports and who will be asked about their career changes prospectively every year
- General population: General population for comparing with previous groups

SUMMARY:
Labor itself can occur spontaneously vaginally, with the help of extraction methods, or via cesarean section. It can also be planned or awaited for the spontaneous onset of uterine contractions. Each method has its advantages and disadvantages regarding potential damage to the pelvic floor and its stability in vaginal delivery or extraction methods, or concerning the stability of the abdominal wall with subsequent wound healing after a cesarean section.

The aim of the study is to retrospectively and prospectively determine the impact of the method of delivery on the performance of female athletes through a questionnaire study. Investigators would like to answer the question of whether cesarean delivery means a later return to training for athletes, whether pregnancy is problematic for female athletes in relation to their BMI, and whether pregnancy often signifies the end of a sports career for female athletes. The questionnaire also includes questions regarding overall women's health-menstrual cycle, incontinence, and mental health of female athletes. Prospectively, the questionnaire will be sent to all female athletes who meet representation limits once a year and for two years after retiring from the national team.

DETAILED DESCRIPTION:
Childbirth and pregnancy are among the most significant moments in a woman's life. The method of delivery is currently a highly debated topic with potential impacts on a woman's future physical and mental health. For elite female athletes, this issue is amplified, as pregnancy and childbirth significantly affect their performance and careers, and it is often necessary to plan pregnancies in consideration of current sporting events and ongoing physical training.

Labor itself can occur spontaneously vaginally, with the help of extraction methods, or via cesarean section. It can also be planned or awaited for the spontaneous onset of uterine contractions. Each method has its advantages and disadvantages regarding potential damage to the pelvic floor and its stability in vaginal delivery or extraction methods, or concerning the stability of the abdominal wall with subsequent wound healing after a cesarean section.

The aim of the study is to retrospectively and prospectively determine the impact of the method of delivery on the performance of female athletes through a questionnaire study. The investigators would like to answer the question of whether cesarean delivery means a later return to training for athletes, whether pregnancy is problematic for female athletes in relation to their BMI, and whether pregnancy often signifies the end of a sports career for female athletes. The questionnaire also includes questions regarding overall women's health-menstrual cycle, incontinence, and mental health of female athletes. Prospectively, the questionnaire will be sent to all female athletes who meet representation limits once a year and for two years after retiring from the national team.

ELIGIBILITY:
Inclusion Criteria:

- Elite female athletes meeting representation limits and included in national teams organized under the Czech Olympic Committee and individual sports federations.

Exclusion Criteria:

- Any male

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Elite female athletes meeting representation limits and included in national teams organized under the Czech Olympic Committee and individual sports federations.
Study Population: General young population for compering with the group of elite athletes which are meeting representation limits and included in national teams organized under the Czech Olympic Committee and individual sports federations.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-16 (Estimated); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Performance | 2 years retrospectively and through study completion, an average of 5 years
  Best score will be used to compare performance of the athletes prior to delivery and after delivery
Performance | 2 years retrospectively and through study completion, an average of 5 years
  Best time will be used to compare performance of the athletes prior to delivery and after delivery
Performance | 2 years retrospectively and through study completion, an average of 5 years
  Most points scored will be used to compare performance of the athletes prior to delivery and after delivery
Placement of athletes during competitions | Prior to delivery and 2 years after the delivery
  Best achievements according to athletes (for example 3rd place on Olympic Games) prior to delivery and after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Antonin Parizek, Prof., MUDr., Study Chair — General Faculty Hospital in Prague
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Ethical approval, Informed consent
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1.6.2025-1.1.2030
Access Criteria: nternational Committee of Medical Journal Editors (ICMJE) and Ethical committee